CLINICAL TRIAL: NCT03072641
Title: Using Probiotics to Reactivate Tumor Suppressor Genes in Colon Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: DuPont Nutrition and Health (Industry)
Responsible Party: Principal Investigator, Yvonne Wettergren, Associate professor, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ALFGBG-542821
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Colon Cancer
Keywords: Probiotics; Epigenetics; Microbiota
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProBion Clinica (Experimental): Probiotic tablets yielding a daily dose of 1.4 x 10 ˄ 10 Bifidobacterium lactis Bl-04 (ATCC SD5219), 7x10 ˄ 9 Lactobacillus acidophilus NCFM (ATCC 700396), and 0.63 g inulin.
  Interventions: Dietary Supplement: ProBion Clinica
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: ProBion Clinica
  Arms: ProBion Clinica

SUMMARY:
The purpose of the study is to determine if probiotic bacteria have a beneficial effect on the colon cancer-associated microbiota and epigenetic alterations in colon cancer. Dietary supplementation consists of two ProBion Clinica tablets, yielding a daily dose of 1.4 x 10 ˄ 10 Bifidobacterium lactis Bl-04 (ATCC SD5219), 7x10 ˄ 9 Lactobacillus acidophilus NCFM (ATCC 700396), and 0.63 g inulin.

ELIGIBILITY:
Inclusion Criteria:

* At least one malignant tumor in the colon

Exclusion Criteria:

* Study subjects with adenomas, or
* who received recent antibiotic therapy or
* consumed probiotics regularly were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in microbiota composition after probiotics use | 8-78 days depending on time elapsed from inclusion to surgical removal of tumor
  The microbiota composition is analysed at baseline and after probiotics use in tissue and faeces samples

SECONDARY OUTCOMES:
Epigenetic changes after probiotics use | 8-78 days depending on time elapsed from inclusion to surgical removal of tumor
  DNA methylation levels are analysed at baseline and after probiotics use in tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne A Wettergren, PhD, Principal Investigator — Dept. of surgery, Sahlgrenska Univ. Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wettergren Y, Rolny P, Lindegren H, Odin E, Rotter Sopasakis V, Keane S, Ejeskar K. Increased MLH1, MGMT, and p16INK4a methylation levels in colon mucosa potentially useful as early risk marker of colon cancer. Mol Cell Oncol. 2025 May 10;12(1):2503069. doi: 10.1080/23723556.2025.2503069. eCollection 2025. PMID 40357388
- [Derived] Keane S, Herring M, Rolny P, Wettergren Y, Ejeskar K. Inflammation suppresses DLG2 expression decreasing inflammasome formation. J Cancer Res Clin Oncol. 2022 Sep;148(9):2295-2311. doi: 10.1007/s00432-022-04029-7. Epub 2022 May 2. PMID 35499706
- [Derived] Hibberd AA, Lyra A, Ouwehand AC, Rolny P, Lindegren H, Cedgard L, Wettergren Y. Intestinal microbiota is altered in patients with colon cancer and modified by probiotic intervention. BMJ Open Gastroenterol. 2017 Jul 3;4(1):e000145. doi: 10.1136/bmjgast-2017-000145. eCollection 2017. PMID 28944067